CLINICAL TRIAL: NCT02909335
Title: De Novo Everolimus Versus Tacrolimus in Combination With Mofetil Mycophenolate and Low Dose Corticosteroids to Reduce Tacrolimus Induced Nephrotoxicity in Liver Transplantation: a Prospective, Multicentric, Randomised Study
Acronym: FOREVER
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 35RC12_8985; 2013-003802-19 (EudraCT Number)
Record Dates: First submitted 2016-09-09; First posted 2016-09-21 (Estimated); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Liver Transplantation
MeSH Terms: interventions — Tacrolimus; Everolimus; Mycophenolic Acid; Prednisolone; Prednisone; Methylprednisolone; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tacrolimus group (Active Comparator): Tacrolimus + mycophenolate mofetil + corticosteroids
  Interventions: Drug: Everolimus; Drug: Mycophenolate mofetil; Drug: Prednisolone, Prednisone or Methylprednisolone
- Everolimus group (Experimental): Everolimus + mycophenolate mofetil + corticosteroids
  Interventions: Drug: Tacrolimus; Drug: Mycophenolate mofetil; Drug: Prednisolone, Prednisone or Methylprednisolone

INTERVENTIONS:
Drug: Tacrolimus — Tacrolimus is administered at an initial dose of 0.040 mg / kg twice a day on Day 5.
  The doses are then adjusted to maintain trough levels :
  * between 6 and 10 ng / ml during the first 2 months,
  * between 5 and 8 ng / ml from the start of the end M3 and M6,
  * and between 4 and 6 ng / ml between the beginning and the end of M7 M12.
  Other Names: Prograf
  Arms: Everolimus group
Drug: Everolimus — Everolimus is administered at an initial dose of 1.5 mg twice a day on Day 5.
  The doses are then adjusted to maintain trough levels:
  * between 6 and 10 ng / ml during the first 2 months,
  * between 5-8 ng / ml from the start of the end M3 and M6,
  * and between 4 and 6 ng / ml between the beginning and the end of M7 M12.
  Other Names: Certican
  Arms: Tacrolimus group
Drug: Mycophenolate mofetil — mycophenolate mofetil is administered similarly in the two groups at the dose of 1.5 g for the first two months and then 1 g twice a day. The doses may be adjusted according to the tolerance of the product.
  Other Names: Cellcept
Drug: Prednisolone, Prednisone or Methylprednisolone — Corticosteroid is similarly administered in both groups between baseline and the end of M6 and adjusted in case of acute rejection
  Other Names: Methylprednisolone: Solumedrol®; Prednisolone: Solupred®; Prednisone: Cortancyl®

SUMMARY:
Tacrolimus is a calcineurin inhibitor. This is the immunosuppression of reference for patients undergoing a first liver transplant. This treatment can prevent graft rejection, but can cause side effects including kidney failure (in 25% after the first year).

Everolimus is an immunosuppressive that effectively prevents acute rejection in heart and kidney transplant recipients. It preserves renal function when it is started soon after the transplant, i.e. before a severe dysfunction is installed.

DETAILED DESCRIPTION:
In the liver transplant, early interruption of calcineurin inhibitors with a quick relay everolimus monotherapy preserves renal function and is associated with a lower acute rejection rate.

We wish to assess whether the introduction of a de novo immunosuppression everolimus under protection of basiliximab induction, mycophenolate mofetil and then low doses of corticosteroids, reduces the nephrotoxicity of immunosuppressive therapy in liver transplant patients, compared to a standard protocol with tacrolimus associated with mycophenolate mofetil and low dose corticosteroids.

ELIGIBILITY:
Pre-transplantation Inclusion Criteria:

* Adults (≥18 years), male or female,
* Patients due to receive a first liver transplant with a full or reduced graft taken from a donor brain-dead beating heart or a related living donor,
* Patients having given a free and informed written consent .

Post-transplantation Inclusion criteria: Patients meeting the following criteria will be included:

* Receiving basiliximab (Simulect)
* Whose immunosuppression regimen from day 5 could immediately consist of either tacrolimus or everolimus, in combination with mycophenolate mofetil and low dose corticosteroids
* With hepatic artery permeable to echo Doppler 4 days after transplant.

Exclusion Criteria:

* History of immunosuppressive therapy,
* Known hypersensitivity to the treatments or macrolides,
* HIV infection
* Autoimmune hepatitis,
* Primary sclerosing cholangitis,
* Programming or realization of a combined transplant,
* Pregnancy or lack of effective contraception,
* Breastfeeding.
* Incompatibility with the donor,
* Thrombosis of the hepatic artery between D0 and D4,
* Non-primary graft function leading to a re-registration on the waiting list.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Worsening of renal function | Between the initiation of treatment (Day 5) and the end (week 48) (censored criterion)
  The main objective of the study is to evaluate, in liver transplanted patients, the benefit in terms of prevention of renal failure, a regimen that includes a de novo introduction of everolimus instead of tacrolimus, in combination with mycophenolate mofetil and low doses of corticosteroids, to the extent that this benefit is not accompanied by an increased risk of graft loss or hepatic artery thrombosis.
  Insofar as the objective of the study is to assess a risk / benefit ratio, the study has two main criteria.
  Worsening renal function is validated before the prolonged decline (found on at least 3 assays carried out at least 3 months apart) over 30% of the creatinine clearance compared to the value at baseline . The date of the first evidence of this worsening of renal function is the date used to calculate the distribution of censored criterion.
Occurrence of graft loss | Between the baseline and the end of the treatment (week 48) (censored criterion
  Graft loss , whatever the cause, or thrombosis of the hepatic artery are recorded between baseline and the end of S48 (censored criterion).

SECONDARY OUTCOMES:
Plasma creatinine | At the end of the treatment (week 48)
Glomerular filtration rate | At the end of the treatment (week 48)
  Glomerular filtration rate calculated following Modification of Diet in Renal Disease (MDRD) formula
Occurrence of mental trouble | Between the baseline and the end of the treatment (week 48) (censored criterion)
  Occurrence of an episode of confusion, agitation or delirium assessed by neurological examination
Occurence of convulsions | Between the baseline and the end of the treatment (week 48) (censored criterion)
  Occurrence of convulsion episodes from baseline to the end of W48 (censored criterion)
Hypertension control | Between the baseline and the end of the treatment (week 48) (censored criterion)
  Occurrence of hypertension requiring the introduction of antihypertensive therapy (censored criterion)
Number of patients with incident diabetes | Between the baseline and the end of the treatment (week 48) (censored criterion)
  Patients presenting development of diabetes requiring the introduction of a hypoglycaemic therapy (censored criterion)
Hypercholesterolemia | Between the baseline and the end of the treatment (week 48) (censored criterion)
  Occurrence of hypercholesterolemia requiring the introduction of lipid-lowering therapy (censored criterion)
Hypertriglyceridemia | Between the baseline and the end of the treatment (week 48) (censored criterion)
  Occurrence of hypertriglyceridemia requiring the introduction of lipid-lowering therapy (censored criterion)
Number of patients with infection | At the end of the treatment (week 48)
  Rate of patients who had at least one infection between baseline and the end of S48 requiring the use of an etiological treatment
Number of everolimus linked adverse events | At the end of the treatment (week 48)
  Rate of patients who had at least one adverse effect of everolimus: ulcer, scar dehiscence, lower limb edema, hyperlipidemia, anemia, leukopenia, thrombocytopenia.
Number of mycophenolate mofetil linked adverse events | At the end of the treatment (week 48)
  Rate of patients who had at least one adverse effect of mycophenolate mofetil: persistent diarrhea, nausea, vomiting, abdominal pain , leukopenia, anemia, thrombocytopenia

CONTACTS AND LOCATIONS:
Overall Officials: Karim BOUDJEMA, MD, PhD, Study Director — CHU Rennes

IPD SHARING:
Plan to Share IPD: No